CLINICAL TRIAL: NCT06751862
Title: The Effect of Simple Carbohydrates on the Development of Non-alcoholic Fatty Liver Disease (FROGLOSA)
Brief Title: The Role of Sugars in Fat Accumulation in the Liver
Acronym: FROGLOSA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for Clinical and Experimental Medicine (Other Government)
Collaborators: Czech Health Research Council (Unknown)
Responsible Party: Principal Investigator, Dita Pajuelo, Principal Investigator, Institute for Clinical and Experimental Medicine
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: AZV NW24J-01-00012
Record Dates: First submitted 2024-11-27; First posted 2024-12-30 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Fatty Liver Disease
Keywords: hepatic fat content; magnetic resonance; fatty liver disease; diet intervention; fructosa; glucosa; sucrosa
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — CD36 Antigens; Glucose; Fructose; Sucrose

STUDY DESIGN:
Intervention Model Description: Part A - Crossover - 2 groups of subjects receive 3 interventions in random order Part B - Single group - the same intervention for all subjects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Part A: male subjects with BMI < 30 kg/m2 (Experimental): Only male subjects with Body Mass Index (BMI) < 30 kg/m2 will be included in this arm.
  The three examinations will be carried out in each subject. The subjects will receive 460 ml of cream (high fat load - 150g of fat in total) with fruit tea sweetened with 50 g of one of the sugars (glucose/fructose/sucrose). Two and four hours later they will receive again fruit tea sweetened with the same sugar as at time 0 h.
  Interventions: Dietary Supplement: 150g of fat with glucose; Dietary Supplement: 150g of fat with fructose; Dietary Supplement: 150g of fat with sucrose
- Part A: male subjects with BMI > 30 kg/m2 (Experimental): Only male subjects with BMI > 30 kg/m2 will be included in this arm. The three examinations will be carried out in each subject. The subjects will receive 460 ml of cream (high fat load - 150g of fat in total) with fruit tea sweetened with 50 g of one of the sugars (glucose/fructose/sucrose). Two and four hours later they will receive again fruit tea sweetened with the same sugar as at time 0 h.
  Interventions: Dietary Supplement: 150g of fat with glucose; Dietary Supplement: 150g of fat with fructose; Dietary Supplement: 150g of fat with sucrose
- Part B: male subjects with steatosis grade 2 (Experimental): Only male subjects with hepatic fat content higher than 6.2% and less than 16.5%, which corresponds to steatosis grade 2, will be included in this arm.
  The subjects will adhere to the diet without fructose for 7 days.
  Interventions: Dietary Supplement: Short-term (7 days) fructose restriction

INTERVENTIONS:
Dietary Supplement: 150g of fat with glucose — The subjects will receive 460 ml of cream (high fat load - 150g of fat in total) with fruit tea sweetened with 50 g of glucose. Two and four hours later they will receive again fruit tea sweetened with the same sugar as at time 0 h. During the day, the subjects will not receive any food and they will be allowed to drink only water or fruit tea.
  Other Names: 460 ml of cream (high fat load - 150g of fat in total) with fruit tea sweetened with 50 g of glucose
  Arms: Part A: male subjects with BMI < 30 kg/m2; Part A: male subjects with BMI > 30 kg/m2
Dietary Supplement: 150g of fat with fructose — Description: The subjects will receive 460 ml of cream (high fat load - 150g of fat in total) with fruit tea sweetened with 50 g of fructose. Two and four hours later they will receive again fruit tea sweetened with the same sugar as at time 0 h. During the day, the subjects will not receive any food and they will be allowed to drink only water or fruit tea.
  Other Names: 460 ml of cream (high fat load - 150g of fat in total) with fruit tea sweetened with 50 g of fructose
  Arms: Part A: male subjects with BMI < 30 kg/m2; Part A: male subjects with BMI > 30 kg/m2
Dietary Supplement: 150g of fat with sucrose — The subjects will receive 460 ml of cream (high fat load - 150g of fat in total) with fruit tea sweetened with 50 g of sucrose. Two and four hours later they will receive again fruit tea sweetened with the same sugar as at time 0 h. During the day, the subjects will not receive any food and they will be allowed to drink only water or fruit tea.
  Other Names: 460 ml of cream (high fat load - 150g of fat in total) with fruit tea sweetened with 50 g of sucrose
  Arms: Part A: male subjects with BMI < 30 kg/m2; Part A: male subjects with BMI > 30 kg/m2
Dietary Supplement: Short-term (7 days) fructose restriction — Subjects will receive a package of glucose and selected foods without fructose to supplement their diet. For seven days they then will adhere to the diet without fructose and keep the detailed dietary record.
  Other Names: 7 days fructose restriction
  Arms: Part B: male subjects with steatosis grade 2

SUMMARY:
This interventional study has 2 parts. In the part A of the project, we will determine how the acute changes in hepatic fat content (HFC) after high-fat load (150 g of fat) are affected by co-administration with three doses of glucose, fructose, and sucrose. HFC in non-obese and obese male volunteers will be measured by magnetic resonance imaging (MRI) and magnetic resonance spectroscopy (MRS) before and at the end of 6-hour intervention. The changes in triglycerides (TG), non-esterified fatty acids (NEFA), insulin and glucose will be also measured throughout the experiments. It can be expected that most of the obese subjects will also have a non-alcoholic fatty liver disease (NAFLD) and we will be therefore able to compare the HFC response between subjects with normal liver fat content and those with steatosis.

Our previous results (doi: 10.26402/jpp.2021.1.05) clearly pointed out that glucose, contrary to fructose, prevents the storage of fat in the liver and that such an effect could be observed even after six hours. In the part B, we will therefore eliminate fructose from the diet of subjects with NAFLD of steatosis grade 2 for seven days - such an intervention will be isocaloric and fructose/sucrose will be replaced by starch or by glucose. The HFC content will be measured again by MRS and MRI after 168 hours. Very low density lipoprotein (VLDL), that transport TG out from the liver, will be isolated before and after intervention from the plasma obtained after overnight fasting. The analysis of lipid profile of the liver fat by MRS and fatty acid profile of TG in VLDL should provide an information on the role of de novo lipogenesis (DNL) in changes of HFC.

In the part A of the project we will aim

* to compare the response of HFC after high-fat load to repeated doses of glucose, fructose, and sucrose (3 x 50 g in two-hour intervals)
* to compare such a response between non-obese and obese-subjects

In the part B of the project we will aim

* to find out whether short-term (7 days) restriction of fructose from the diet will decrease HFC in subjects with NAFLD
* to find out whether such an intervention affects fatty acid profile of hepatic TG evaluated by MRS and by fatty acid profile of TG in VLDL - in this way we can estimate whether DNL is suppressed after fructose withdrawal
* to further corroborate such an aim, we will also compare the fatty acid profile of plasma NEFA and that of TG in VLDL

DETAILED DESCRIPTION:
1. INTRODUCTION Non-alcoholic fatty liver disease (NAFLD) is currently the leading cause of chronic liver disease, it affects approximately one-quarter of the global population and the incidence of the disease is still rising (doi: 10.1210/endrev/bnz009). The occurrence of NAFLD is tightly associated with the obesity, insulin resistance and/or type 2 diabetes (doi: 10.7759/cureus.20776). Some authors even consider NAFLD to be hepatic manifestation of metabolic syndrome or even the precursor of metabolic syndrome development (doi: 10.1016/j.dld.2014.09.020).

   The growing incidence of NAFLD has been attributed to sedentary life-style, energy intake inadequate to energy expenditure and also to increased intake of simple carbohydrates (added sugars), and specifically, increased intake of fructose (both as a part of sucrose molecule and also, especially in the United States (US), as a component of high-fructose corn syrup (HFCS)). Over the last decades, a number of papers have been presented which have shown a link between increased consumption of added sugars (especially of fructose) and the obesity and insulin resistance pandemic (doi: 10.1097/MOL.0b013e3283613bca, doi: 10.1007/s00394-018-1711-4, doi: 10.1016/j.nut.2013.08.014).

   However, recent meta-analyses have not supported the role of increased added sugar or fructose intake in development of obesity, insulin resistance, metabolic syndrome and type 2 diabetes (doi: 10.1017/S0954422414000067, doi: 10.1007/s00394-016-1345-3). They rather suggest that the added sugars are detrimental if associated with inadequately increased energy intake. It was even suggested that increased fructose/added sugars consumption may be a marker of unhealthy life-style. On the other hand, not so many data are available with respect to the role of added sugars and, specifically, fructose, in the development of fatty liver.

   This may be due to the fact that the metabolism of glucose and fructose metabolism in the liver is fundamentally different (doi: 10.1016/j.jada.2010.06.008, doi: 10.3390/nu9091026, doi: 10.1016/j.clnu.2020.12.022). Contrary to glucose, which is largely metabolized by extrahepatic tissues, most of fructose is directly uptaken and metabolized by the liver. Moreover, phosphorylation of fructose to fructose-1-phosphate catalyzed by fructokinase/ketohexokinase is not under any feedback control and results in uncontrolled production of trioso-3-phosphates. These can enter gluconeogenesis pathway and be further used to replete glycogen (in state of glycogen depletion) but they can also provide a substrate for de novo lipogenesis (DNL) and, at the same time, inhibit fatty acid oxidation. Fructose seems to be also a potent activator of carbohydrate-responsive element-binding protein (ChREBP) regulatory pathway that together with sterol regulatory element-binding protein (SREBP) promotes DNL in the liver.

   Importantly, in spite of the fact that fatty acids released from adiposse tissue are the major source of the liver fat, the contribution of DNL to liver fat accumulation significantly increases specifically in patients with NAFLD (doi: 10.1172/JCI23621, doi: 10.1053/j.gastro.2013.11.049).

   Studies looking at the effect of fructose consumption on hepatic fat content (HFC) have not reach a clear conclusion. In healthy subjects, fructose administration under isocaloric conditions does not seem to have any impact on HFC (doi: 10.1093/ajcn/84.6.1374, doi: 10.1093/ajcn/nqz271). Fat accumulated in the livers of healthy subjects only when exposed to a hypercaloric high-fructose diet (doi: 10.3945/ajcn.2008.27336). On the contrary, abdominally obese men accumulated more fat in the liver even on an isocaloric high-fructose diet (doi: 10.1111/joim.12632). Interestingly, in the study comparing a high-glucose and high-fructose diet under both iso- and hypercaloric conditions, overweight men accumulated liver fat in the liver only under hypercaloric conditions but no difference in the effect on HFC was found between glucose and fructose (doi: 10.1053/j.gastro.2013.07.012).
2. PILOT DATA Glucose and fructose can have different effects in the accumulation of fat in the liver which we have demonstrated in our studies of acute changes of HFC after nutrient administration (doi: 10.1093/ajcn/nqy386, doi: 10.26402/jpp.2021.1.05). In these studies we developed and introduced a functional test that allowed us to monitor acute changes in hepatic fat after a challenge with high-fat and/or simple carbohydrate load. In the test, the 150 g of fat is administered to subjects at the beginning of experiment, whereas carbohydrates (50 g of fructose or glucose) are administered every 2 hours to efficiently suppress the lipolysis in adipose tissue as documented by suppression of non-esterified fatty acids (NEFA) concentration (doi: 10.1093/ajcn/nqy386). In this way we can limit the impact of fatty acids from the adipose tissue on accumulation of hepatic fat and the resulting changes should be explained by contribution of dietary fat or DNL.

   Importantly, in this model we have shown that 6 hours after consumption of 150 g of fat (cream), HFC increases in both healthy non-obese subjects with normal fat content (doi: 10.1093/ajcn/nqy386) and also in non-obese subjects with hepatosteatosis (doi: 10.26402/jpp.2021.1.05). Liver fat increases also when fructose is co-administered with fat. On the contrary, glucose co-administration with fat prevents such an increase in HFC (doi: 10.1093/ajcn/nqy386, doi: 10.26402/jpp.2021.1.05).
3. THE RATIONALE OF THE PROJECT The added sugars represent more than 12% of daily energy intake. Their role in accumulation of liver fat has been studied so far with pure glucose or pure fructose. However, in real life people do not consume pure glucose or fructose, they consume fructose together with glucose both as a part of sucrose or in high-fructose corn syrup. It is not entirely clear how the hepatic fat content will respond to the mixture of both sugars. The question how concurrent consumption of both hexoses affect the accumulation of fat in the liver may be of great practical significance and answering this question might greatly contribute to the modification of dietary recommendations for NAFLD treatment.

   Importantly, as we were unable to demonstrate the difference between the response of HFC to glucose and fructose administration in non-obese non-diabetic subjects (doi: 10.26402/jpp.2021.1.05), it would be preferable to study the acute effects of these three sugars on HFC after their co-administration with high-fat load.

   The number of studies clearly documented adverse effects of excessive fructose consumption on metabolic health. On the other hand, if fructose does harm human health, it would be important to know whether fructose restriction has an effect on HFC. Indeed, fructose restriction led to a significant reduction in liver fat after 9 days in obese children (doi: 10.1053/j.gastro.2017.05.043) and after 6 weeks in obese individuals (doi: 10.1093/ajcn/nqaa332). Based on our previous results, it can be hypothesized that eliminating fructose from the diet and replacing it by starch or glucose should effectively suppress hepatic fat content even in a few days.
4. HYPOTHESES

   Two principal hypotheses will be tested:
   * The increase of hepatic fat content after high-fat load is blunted by glucose but not fructose neither sucrose (Part A of the project).
   * The short-term (7 days) dietary fructose restriction results in a decrease of hepatic fat content (Part B of the project)
5. EXPERIMENTAL DESIGN Part A The design of this part of the study will be the same as that in our previous studies (doi: 10.1093/ajcn/nqy386, doi: 10.26402/jpp.2021.1.05) except that only two measurements of hepatic fat content (HFC) by magnetic resonance spectroscopy (MRS) will be carried out during each experiment. The three examinations lasting approximately 8 hours will be carried out in each subject in the study. First, hepatic fat content (HFC) will be measured using MRS (30-45 mins). The cannula will be then inserted into the antecubital vein and the first blood draw will be carried out. The subjects will then receive 460 ml of cream (high fat load - 150g of fat in total) with fruit tea sweetened with 50 g of one of the sugars (glucose/fructose/sucrose). Two and four hours later they will receive again fruit tea sweetened with the same sugar as at time 0 h. The blood for biochemical analyses will be then taken at 0.5, 1, 2 (before tea), 2.5, 3, 4 (before tea), 4.5, 5 and 6 hours. During the day, the subjects will not receive any food and they will be allowed to drink only water or fruit tea. The measurement of hepatic fat content will be repeated at time 6 hours. During magnetic resonance (MR) examination the volume of visceral fat will be also measured and body composition will be determined. The order of examinations will be randomized and they will be carried out in at least two-week intervals.

   Subjects: Two groups of male volunteers will be studied in this part of the project - 15 nonobese subjects (Body Mass Index (BMI) < 30 kg/m2) and 15 obese subjects (BMI ˃ 30 kg/m2). The subjects will be 18 - 70 years old and groups will be age-matched. Based on our previous studies with healthy male subjects the number of 13 subjects in one group should be sufficient to detect 10 ± 10% increment in HFC after the fat load at α = 0.05 (two-tailed paired t-test) and β = 0.10. The slightly higher number per group covers the risks associated with the exclusion or withdrawal of some subjects during the study.

   The exclusion criteria for both groups will be diabetes mellitus (fasting glucose above 7 mmol/l, 2-hour glucose after oGTT ˃ 11.1 mmol/l, or antidiabetic treatment) or other serious illnesses (cardiovascular disease, cancer, etc.), alcohol consumption ˃ 30 g/day, fructose intolerance, use of drugs affecting lipid metabolism and intolerance of MR examination (claustrophobia, metal implants, etc.). Before the entry into the study, subjects will sign the informed consents with participation in the study and genetic tests and before each experiment they will sign the informed consent with MR examination.

   Part B Subjects selected for this part of the study will first complete a detailed three-day dietary record allowing us to quantify their fructose consumption among other things. They will then be instructed in detail how to change their diet to eliminate fructose and receive these recommendations also in writing. On the first day of the seven-day dietary intervention, they will have fasting blood drawn and then the hepatic fat content will be measured by MRS. After that they will receive a package of glucose and selected foods without fructose to supplement their diet. For seven days they then will adhere to the diet without fructose and keep the detailed dietary record. On the last day of the intervention, they will have fasting blood drawn and HFC measured by MRS again (after 168 hours exactly).

   Subjects: Fifteen subjects 18 to 70 years old will be included in the study. Similarly as in Part A, such a number of subjects is slightly higher than 13 - a number sufficient to detect 10 ± 10% decrease in HFC at α = 0.05 (two-tailed paired t-test) and β = 0.10.

   To be included, the hepatic fat content in the subjects must be higher than 6.2% and less than 16.5% which corresponds to steatosis grade 2 (doi: 10.1007/s10334-011-0264-9). The participants of Part A of the study meeting this criterion can be also included in Part B. The exclusion criteria will be the same as in Part A. Before the entry into the study, subjects will sign the informed consents with participation in the study and genetic tests and before each experiment they will sign the informed consent with MR examination.
6. METHODS MR spectroscopy (MRS). Standard single voxel spectroscopy sequence with breath holding (3 Tesla VIDA Siemens magnetic resonance (MR) system equipped with multi-channel surface body coil) will be used to measure hepatic fat content (HFC). MR images in three anatomical orientations will be used to set the volume of interest of 40x30x25 mm. The correction of signal intensities to T2 relaxation will be done.

   To get information about lipid profile of the liver triglycerides (TG) the MRS spectra will be analyzed as described earlier (doi: 10.3390/metabo11090625.).

   HISTO MR imaging (MRI). Proton Density Fat Fraction (PDFF) imaging will be measured by HISTO Siemens protocol approved by Food and Drug Administration (FDA). It includes spectroscopic, Dixon and multiecho Dixon sequences.

   Data evaluation. MR spectra will be evaluated using the LCModel (doi: 10.1002/nbm.698) and percentage of HFC assessed by MRS will be calculated according to Longo (doi: 10.1002/jmri.1880050311).

   Visceral fat content measurement by MR imaging. The content of visceral fat will be measured by turbo spin echo sequence before or after PDFF measurement. To evaluate the volume of visceral and subcutaneous fat software written in MATLAB will be used. To reduce the impact of the operator, visceral fat areas will be evaluated by two independent experts.

   Body composition. The body composition during the screening will be determined using InBody.

   Biochemical analysis. The blood will be collected into tubes containing all necessary inhibitors, immediately placed on the ice and centrifuged to collect plasma within 15 min. Glucose, triglyceride (TG), non-esterified fatty acids (NEFA), insulin, and β-hydroxybutyrate will be measured in all the samples obtained in the study. All the necessary biochemical, Radioimmunoassay (RIA) and enzyme-linked immunosorbent assay (ELISA) methods for determination of these parameters are currently in use in the laboratories of applicants.

   Lipidomics. The VLDL will be isolated by ultracentrifugation, and the analysis of fatty acid profile of VLDL-triglycerides and plasma free fatty acids will be carried out by liquid chromatography - mass spectrometry (LC-MS) in Metabolomics department of Institute of Physiology, Czech Academy of Sciences (paid service).

   Genetics. The polymorphisms of genes (PNPLA, TM6SF2, and others) known to affect accumulation of liver fat will be determined.

   Statistics. Statistical data analysis and correlations will be performed with PRISM 9.1 or JMP software.
7. TIME SCHEDULE OF THE PROJECT 2024: Part A: Preparation of study protocols, search and screening of subjects, start of the study examinations in first subjects - approximately 20 whole-day examinations will be carried out of 90 examinations total (3 examinations per each of 30 subjects). The number of subjects that can be studied is limited by the availability of MR tomograph for research studies (1 day a week) and complexity of examinations. Basic biochemical analyses will be carried out continuously but all the samples from each subject (30 total) will be stored at -80°C and analyzed simultaneously.

Part B: Preparation of study protocols and dietary records that can be used for quantification of fructose consumption. Search and screening of subjects.

2025: Part A: Screening of subjects, study examinations - min. 30 whole-day examinations will be carried out. Continuation of biochemical analyses.

Part B: Screening of subjects (subjects with hepatosteatosis studied in Part A can be also included in Part B). Dietary intervention experiments (approx. n=20) in approx. 10 subjects (1 subject a week can be intervened, including MR examination and overnight isolation of VLDL on the first and the last day of intervention). Biochemical analyses.

2026: Part A: Screening of subjects, study examinations - min. 30 whole-day examinations will be carried out. Continuation of biochemical analyses. Start of intensive data analysis.

Part B: Screening of subjects. Dietary intervention experiments (n = 10) in remaining subjects on the first and the last day of intervention. Biochemical analyses. Specialized biochemical analyses (for example, ELISA for fibroblast rowth factor 19 (FGF-19), selected hepatokines or other proteins that can be involved in regulation of de novo lipogenesis) and lipidomic analysis of fatty acid profile in free fatty acid (FFA) pool and TG in VLDL. Analysis of the data and publication of results.

2027: Part A: Study examinations in remaining subjects - max. 10 whole-day examinations will be carried out. Continuation of routine biochemical analyses. Specialized biochemical analyses (see above). Analysis of the data and publication of results.

Part B: Final analysis of the data and publication of results.

8. ANTICIPATED RESULTS This project will provide new insights into the mechanisms by which simple carbohydrates affect the accumulation of liver fat. Of particular importance will be comparison the role of fructose and glucose (which are intensively studied but not used by population) and that of sucrose, the sugar generally used to sweeten by the whole population. Moreover, the experiment with fructose restriction from the diet should determine whether such an intervention can be useful for treatment of hepatosteatosis. On the whole, both parts of the projects should provide the results that can be implemented in practical dietary recommendations and improve the strategies for management of NAFLD.

ELIGIBILITY:
Part A

Inclusion Criteria:

* male volunteers - 15 nonobese subjects (Body Mass Index (BMI) < 30 kg/m2) and 15 obese subjects (BMI ˃ 30 kg/m2)
* 18 - 70 years old

Exclusion Criteria:

* diabetes mellitus (fasting glucose above 7 mmol/l, 2-hour glucose after oGTT above 11.1 mmol/l, or antidiabetic treatment)
* other serious illnesses (cardiovascular disease, cancer, etc.)
* alcohol consumption ˃ 30 g/day
* fructose intolerance
* use of drugs affecting lipid metabolism

Part B

Inclusion Criteria:

* male volunteers with hepatic fat content higher than 6.2% and less than 16.5%, which corresponds to steatosis grade 2 (S2)
* 18 - 70 years old

Exclusion Criteria:

* diabetes mellitus (fasting glucose above 7 mmol/l, 2-hour glucose after oGTT above 11.1 mmol/l, or antidiabetic treatment)
* other serious illnesses (cardiovascular disease, cancer, etc.)
* alcohol consumption ˃ 30 g/day
* use of drugs affecting lipid metabolism
* intolerance of MR examination (claustrophobia, metal implants, etc.).

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
The comparison of the increment of hepatic fat content after high-fat load to repeated doses of glucose, fructose, and sucrose | Three one-day measurements (8 hours) 2 weeks apart, from enrollment to the last intervention at aprox. 8 weeks
  The three examinations lasting approx. 8 hours will be carried out in each subject in the study. First, hepatic fat content will be measured using magnetic resonance imaging and magnetic resonance spectroscopy. The cannula will be then inserted into the antecubital vein and the first blood draw will be carried out. The subjects will then receive 460 ml of cream with fruit tea sweetened with 50 g of one of the sugars (glucose/fructose/sucrose). Two and four hours later they will receive again fruit tea sweetened with the same sugar as at time 0 h. The blood for biochemical analyses will be then taken at 0.5, 1, 2 (before tea), 2.5, 3, 4 (before tea), 4.5, 5 and 6 hours. The measurement of hepatic fat content will be repeated at time 6 hours. During MR examination the volume of visceral fat will be also measured and body composition will be determined. The order of examinations will be randomized and they will be carried out in at least two-week intervals.
The comparison of the increment of HFC after high-fat load with repeated doses of simple sugar between non-obese and obese-subjects | Three one-day measurements (8 hours) 2 weeks apart, from enrollment to the last intervention at aprox. 8 weeks
  The three examinations lasting approx. 8 hours will be carried out in each subject in the study. First, hepatic fat content will be measured using magnetic resonance imaging and magnetic resonance spectroscopy. The cannula will be then inserted into the antecubital vein and the first blood draw will be carried out. The subjects will then receive 460 ml of cream with fruit tea sweetened with 50 g of one of the sugars (glucose/fructose/sucrose). Two and four hours later they will receive again fruit tea sweetened with the same sugar as at time 0 h. The blood for biochemical analyses will be then taken at 0.5, 1, 2 (before tea), 2.5, 3, 4 (before tea), 4.5, 5 and 6 hours. The measurement of hepatic fat content will be repeated at time 6 hours. During MR examination the volume of visceral fat will be also measured and body composition will be determined. The order of examinations will be randomized and they will be carried out in at least two-week intervals.
The comparison of hepatic fat content values after short-term (7 days) restriction of fructose from the diet in subjects with fatty liver | From the beginning to the end of the intervention at 7 days
  The fructose will be eliminated from the diet of subjects with fatty liver of steatosis grade 2 (S2) for seven days - such an intervention will be isocaloric and fructose/sucrose will be replaced by starch or by glucose. On the first day of the seven-day dietary intervention, the hepatic fat content (HFC) will be measured by magnetic resonance spectroscopy (MRS). After that they will receive a package of glucose and selected foods without fructose to supplement their diet. For seven days they then will adhere to the diet without fructose and keep the detailed dietary record. On the last day of the intervention, HFC will be measured by MRS again (after 168 hours exactly).
Change of hepatic fatty acid profile after short-term restriction of fructose | From enrollment to the analysis at 2 years
  The hepatic fatty acid profile will be calculated from magnetic resonance spectroscopy (MRS) and magnetic resonance imaging (MRI) data before and after short-term restriction of fructose.
Change of fatty acid profile of triglycerides in very low-density lipoproteins after short-term restriction of fructose | From enrollment to the analysis at 2 years
  Very low-density lipoproteins (VLDL) will be isolated by ultracentrifugation and the fatty acid profile of VLDL-triglycerides will be measured by liquid chromatography - mass spectrometry (LC-MS) in Metabolomics department of Institute of Physiology, Czech Academy of Sciences (paid service). Fatty acid profile of VLDL-triglycerides will be then compared before and after short-term restriction of fructose.
Change of fatty acid profile of plasma non-esterified fatty acids after short-term restriction of fructose | From enrollment to the analysis at aprox. 30 months
  Plasma free fatty acids will be carried out by liquid chromatography - mass spectrometry (LC-MS) in Metabolomics department of Institute of Physiology, Czech Academy of Sciences (paid service). Plasma free fatty acid profile will be then compared before and after short-term restriction of fructose.

SECONDARY OUTCOMES:
Frequency of polymorphisms of PNPLA3, TM6SF2, and other genes affecting accumulation of liver fat in each study group | From enrollment to the analysis at aprox. 24 months
  The frequency of gene polymorphisms (PNPLA3, TM6SF2, and others) will be compared between the group with BMI < 30 kg/m2 and the group with BMI > 30 kg/m2 .

CONTACTS AND LOCATIONS:
Overall Officials: Dita Pajuelo, PhD, Principal Investigator — Institute for Clinical and Experimental Medicine
Locations (1):
- Institute for Clinical and Experimental Medicine, Prague, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: No
However, the anonymized data that support the findings of this study might be available from the corresponding author upon reasonable request.

REFERENCES:
- [Background] Burian M, Hajek M, Sedivy P, Mikova I, Trunecka P, Dezortova M. Lipid Profile and Hepatic Fat Content Measured by 1H MR Spectroscopy in Patients before and after Liver Transplantation. Metabolites. 2021 Sep 15;11(9):625. doi: 10.3390/metabo11090625. PMID 34564441
- [Background] Hajek M, Dezortova M, Wagnerova D, Skoch A, Voska L, Hejlova I, Trunecka P. MR spectroscopy as a tool for in vivo determination of steatosis in liver transplant recipients. MAGMA. 2011 Oct;24(5):297-304. doi: 10.1007/s10334-011-0264-9. Epub 2011 Jul 10. PMID 21744232
- [Background] Kovar J, Dusilova T, Sedivy P, Bruha R, Gottfriedova H, Pavlikova P, Pitha J, Smid V, Drobny M, Dezortova M, Hajek M. Acute responses of hepatic fat content to consuming fat, glucose and fructose alone and in combination in non-obese non-diabetic individuals with non-alcoholic fatty liver disease. J Physiol Pharmacol. 2021 Feb;72(1). doi: 10.26402/jpp.2021.1.05. Epub 2021 Jun 3. PMID 34099584
- [Background] Dusilova T, Kovar J, Drobny M, Sedivy P, Dezortova M, Poledne R, Zemankova K, Hajek M. Different acute effects of fructose and glucose administration on hepatic fat content. Am J Clin Nutr. 2019 Jun 1;109(6):1519-1526. doi: 10.1093/ajcn/nqy386. PMID 31136656